CLINICAL TRIAL: NCT00934336
Title: Importance in Type 1 Diabetes Patients of an Optimized Control of Post-Prandial Glycaemia on Oxidant Stress Prevention
Acronym: ITOPOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2007-A01036-47
Record Dates: First submitted 2009-07-07; First posted 2009-07-08 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2011-02

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- preprandial injection (Experimental): pre-prandial injection of an ultra-fast-acting analog during 3 months, then post-prandial injection of an ultra-fast-acting analog during 3 other months.
  Interventions: Other: Therapeutic and preventive strategies
- post-prandial injection (Experimental): post-prandial injection of an ultra-fast-acting analog during 3 months then pre-prandial injection of an ultra-fast-acting analog during 3 other months.
  Interventions: Other: Therapeutic and preventive strategies

INTERVENTIONS:
Other: Therapeutic and preventive strategies — These results may help us to define a post prandial insulin treatment regimen (which is more flexible as regards meals) or a pre prandial insulin treatment regimen (less flexible for meals but maybe less harmful in terms of limitation of oxidative stress).
  Arms: preprandial injection
Other: Therapeutic and preventive strategies — These results may help us to define a post prandial insulin treatment regimen (which is more flexible as regards meals) or a pre prandial insulin treatment regimen (less flexible for meals but maybe less harmful in terms of limitation of oxidative stress).
  Arms: post-prandial injection

SUMMARY:
The aim of this study is to determine whether postprandial hyperglycaemia plays an important role in oxidative stress phenomena and influences their harmful effects on the arterial wall.

25 type 1 diabetic patients practicing FIT and with an HbA1c value of 8 percent or less at the beginning of the study will be recruited. The 25 control subjects will be recruited after the patients, so that they can be paired by age and sex.

Patients will be randomized via an alternative cross over study design for 2 periods of 3 months, i.e. preprandial or postprandial injection of an ultra fast acting analog. During the 6 months of the study, slow acting analog doses will be adjusted on the basis of basal glycaemia values. The fast acting analog doses will be adjusted on the basis of an optimized algorithm available on each patient's PDA phone electronic diary.

Blood and urine samples will be collected at M0, M3 and M6 to evaluate the stress oxidant grade and its consequence on atherogenesis:

Oxidative Stress evaluation: plasma parameters (lipid peroxide derivatives, semicarbazide sensitive oxidase amine activity), erythrocyte and leukocyte cell parameters (reduced and oxidised glutathion, dismutase superoxide activity (SOD) Cu and Mn dependent, glutathion peroxidase, and catalase), urinary parameters (isoprostane F2) Evaluation of consequences of oxidative stress on atherogenesis processes: inflammatory parameters (CRP, TNFa, IL 6), adhesion molecules (VCAM 1, ICAM 1, P selectine), adipokines (leptine, resistine, adiponectine), coagulation factors (PAI 1), platelet and endothelial microparticles, The pre and postprandial glycaemic stability of each patient will be monitored using PDA phone systems, and HbA1c will be measured at M0, M3 and M6.

Expected results and outcomes:

It is important to know if, in patients with comparable glycaemic stability, these two insulin treatment regimens are associated with significant differences in oxidative stress and anti oxidant defenses.

These results may help us to define a postprandial insulin treatment regimen (which is more flexible as regards meals) or a preprandial insulin treatment regimen (less flexible for meals but maybe less harmful in terms of limitation of oxidative stress).

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes
* treaties by basal / bolus with a ultra rapid analogue or a pump with a ultra rapid analogue
* Adults between 18 and 50 years old
* Patients practicing FIT
* Written informed consent obtained prior to enrollment in the study
* HbA1c ≤ 8%

Exclusion Criteria:

* Diabetes other than DT1
* Complications: coronary or peripheral arteriopathy
* Pathologies being able to interfere with the study: HTA, dyslipidemia, nicotinism, inflammatory , cancerous pathology…
* Psychiatric pathologies incompatible with the study
* Pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2008-11; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Assay of isoprostane-F2, an indicator of lipid peroxidase derivative production, in the 24 hour urine | T0, T3 months, T6 months

CONTACTS AND LOCATIONS:
Overall Officials: FEVE Bruno, MD PH, Study Chair — Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète; CHARPENTIER Guillaume, PH, Principal Investigator — CH Sud Francilien
Locations (1):
- CH sud francilien, Corbeil-Essonnes, France